CLINICAL TRIAL: NCT01479374
Title: A Multi-Center, Randomized, Double-Masked, Vehicle and Active Controlled, Parallel-Group Efficacy and Safety Study of AL-4943A Ophthalmic Solution, 0.77% in Patients With Allergic Conjunctivitis Using the Conjunctival Allergen Challenge (CAC) Model
Brief Title: Efficacy and Safety of AL-4943A Ophthalmic Solution in Patients With Allergic Conjunctivitis Using the Conjunctival Allergen Challenge (CAC) Model
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C-10-126
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Results first posted 2013-05-23 (Estimated); Last update posted 2013-06-04 (Estimated); Status verified 2013-05

CONDITIONS: Allergic Conjunctivitis
Keywords: Allergic Conjunctivitis; Ocular Allergy
MeSH Terms: conditions — Conjunctivitis, Allergic | interventions — Olopatadine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- AL-4943A (Experimental): AL-4943A ophthalmic solution, 1 drop to each eye, 3 nonconsecutive days
  Interventions: Drug: AL-4943A ophthalmic solution
- Vehicle (Placebo Comparator): AL-4943A vehicle, 1 drop to each eye, 3 nonconsecutive days
  Interventions: Drug: AL-4943A vehicle
- Pataday (Active Comparator): Olopatadine hydrochloride ophthalmic solution, 0.2%, 1 drop to each eye, 3 nonconsecutive days
  Interventions: Drug: Olopatadine hydrochloride ophthalmic solution, 0.2%

INTERVENTIONS:
Drug: AL-4943A ophthalmic solution
  Arms: AL-4943A
Drug: AL-4943A vehicle — Inactive ingredients used as placebo
  Arms: Vehicle
Drug: Olopatadine hydrochloride ophthalmic solution, 0.2%
  Other Names: PATADAY®
  Arms: Pataday

SUMMARY:
The purpose of this study was to assess the safety and efficacy of AL-4943A ophthalmic solution for the treatment of ocular itching associated with allergic conjunctivitis using the Conjunctival Allergen Challenge (CAC) model.

DETAILED DESCRIPTION:
This study consisted of 5 Visits. Eligible patients underwent allergy testing using the Conjunctival Allergen Challenge (CAC) model, which reproduces the signs and symptoms of Seasonal Allergic Conjunctivitis by replicating the natural disease process. Patients demonstrating a positive reaction to the CAC at Visit 1 (screening) and Visit 2 (confirmatory) were randomized to treatment at Visit 3 (Day 0). The test article was instilled at Visit 3, with treatment efficacy CAC performed at 24 hours duration of action. The test article was instilled again at Visit 4 (Day 14), with treatment efficacy CAC performed at 16 hours duration of action. The test article was instilled a final time at Visit 5 (Day 21), with treatment efficacy performed at onset of action.

ELIGIBILITY:
Inclusion Criteria:

* Able to be dosed in both eyes, able and willing to make the required study visits and to follow instructions.
* Diagnostic skin test indicative of allergy for cat hair, cat dander, grasses, ragweed, dust mite, dog dander, cockroach and/or trees within 24 months of Visit 1.
* History of seasonal or perennial allergic conjunctivitis for at least 1 year prior to Visit 1.
* Positive bilateral CAC response at Visit 1 and Visit 2.
* Willing to discontinue contact lens wear for at least 72 hours prior to Visit 1 and throughout the study.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Known history or presence of persistent dry eye syndrome, or currently requiring frequent use (> 4 days per week) of artificial tears, gels or lubricants, presence of punctal plugs, use of Restasis®, or topical ocular corticosteroids for dryness of eyes.
* Presence of active blepharitis, active meibomian gland dysfunction, active rosacea affecting the ocular adnexa, follicular conjunctivitis, iritis, preauricular lymphadenopathy, ocular irritation not due to ocular allergy, or any other clinically significant ophthalmic abnormality that may affect the study outcomes.
* Presumed or actual ocular infection (bacterial, viral or fungal) or history of ocular herpes in either eye as determined by patient history and/or examination within 30 days of Visit 1.
* Presence of any chronic ocular degenerative condition or active intra-ocular inflammation in either eye that in the opinion of the Investigator is likely to advance/worsen during the time course of the study.
* Any contraindications or hypersensitivities to the use of the study medication or their components.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 397 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Abhijit Narvekar, MS, MBBS, Study Director — Alcon Research

REFERENCES:
- [Derived] Carr W, Schaeffer J, Donnenfeld E. Treating allergic conjunctivitis: A once-daily medication that provides 24-hour symptom relief. Allergy Rhinol (Providence). 2016 Jan;7(2):107-14. doi: 10.2500/ar.2016.7.0158. Epub 2016 Jul 26. PMID 27466061

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from three US study centers.
Pre-assignment Details: Of the 397 enrolled, 195 subjects did not qualify for treatment and were exited without exposure to product. Participant flow and baseline characteristics are presented for the 202 subjects qualifying for treatment and randomized 1:1:1 to receive AL-4943A, Vehicle, or Pataday.
Period: Overall Study
Arm/Group | AL-4943A | Vehicle | Pataday
Started | 66 | 68 | 68
Completed | 63 | 60 | 63
Not Completed | 3 | 8 | 5
Not completed — Adverse Event | 2 | 1 | 0
Not completed — Lost to Follow-up | 1 | 2 | 0
Not completed — Decision Unrelated to Adverse Event | 0 | 1 | 0
Not completed — Other | 0 | 4 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AL-4943A | Vehicle | Pataday | Total
Number analyzed (Participants) | 66 | 68 | 68 | 202
Age, Customized [Number; unit: participants]
  18 to 64 years | 64 | 66 | 66 | 196
  >=65 years | 2 | 2 | 2 | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 39 | 42 | 124
  Male | 23 | 29 | 26 | 78
Region of Enrollment [Number; unit: participants]
  United States | 66 | 68 | 68 | 202

OUTCOME MEASURES:

1. Primary Outcome: Mean Ocular Itching at Onset of Action
Description: A treatment efficacy CAC was performed 27 minutes after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=incapacitating itch). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, and 7 minute timepoints, post-CAC on Day 21 of receiving treatment
Population: Intent to treat (ITT). The analysis population included all randomized patients who received treatment and had post CAC data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 63 | 60 | 63
Units on a scale
  3 min post-CAC | 0.4 (0.7) | 1.9 (1.1) | 0.4 (0.6)
  5 min post-CAC | 0.6 (0.8) | 2.1 (1.1) | 0.7 (0.7)
  7 min post-CAC | 0.5 (0.7) | 2.0 (1.1) | 0.7 (0.8)

2. Primary Outcome: Mean Ocular Itching at 16 Hours Duration of Action
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=incapacitating itch). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, and 7 minute timepoints, post-CAC on Day 14 of receiving treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 65 | 65 | 65
Units on a scale
  3 min post-CAC | 0.7 (0.7) | 2.2 (0.9) | 0.9 (0.8)
  5 min post-CAC | 0.8 (0.8) | 2.3 (0.9) | 1.1 (1.0)
  7 min post-CAC | 0.8 (0.9) | 2.1 (0.9) | 1.0 (0.9)

3. Secondary Outcome: Mean Conjunctival Redness at Onset of Action
Description: A treatment efficacy CAC was performed 27 minutes after drop instillation. Conjunctival redness was assessed by the investigator on a 0-4 scale (0=none to 4=extremely severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, and 20 minute timepoints, post-CAC on Day 21 of receiving treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 63 | 60 | 63
Units on a scale
  7 min post-CAC | 0.8 (0.7) | 2.1 (0.7) | 1.3 (0.8)
  15 min post-CAC | 1.1 (0.9) | 2.3 (0.6) | 1.9 (0.8)
  20 min post-CAC | 1.1 (0.8) | 2.3 (0.7) | 1.9 (0.8)

4. Secondary Outcome: Mean Conjunctival Redness at 16 Hours Duration of Action
Description: A treatment efficacy CAC was performed 16 hours after drop instillation. Conjunctival redness was assessed by the investigator on a 0-4 scale (0=none to 4=extremely severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, and 20 minute timepoints, post-CAC on Day 14 of receiving treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 65 | 65 | 65
Units on a scale
  7 min post-CAC | 1.3 (0.8) | 1.8 (0.8) | 1.6 (0.7)
  15 min post-CAC | 1.5 (0.8) | 1.9 (0.8) | 1.9 (0.7)
  20 min post-CAC | 1.5 (0.8) | 1.9 (0.9) | 1.9 (0.7)

5. Secondary Outcome: Mean Total Redness at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Total redness (0-12) is defined as the sum of ciliary redness (0-4 scale, from 0=none to 4=extremely severe), conjunctival redness (0-4 scale, from 0=none to 4=extremely severe), and episcleral redness (0-4 scale, from 0=none to 4=extremely severe). Average of total redness score over both eyes was analyzed.
Time Frame: 7, 15, and 20 minute timepoints, post-CAC on Day 1 of receiving treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 66 | 68 | 66
Units on a scale
  7 min post-CAC | 4.1 (2.6) | 6.1 (2.3) | 5.4 (2.4)
  15 min post-CAC | 5.0 (2.9) | 6.7 (2.3) | 6.2 (2.3)
  20 min post-CAC | 5.4 (2.9) | 6.6 (2.6) | 6.3 (2.3)

6. Secondary Outcome: Mean Ocular Itching at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Ocular itching was assessed by the patient on a 0-4 scale (0=none to 4=incapacitating itch). Average of ocular itching score over both eyes was analyzed.
Time Frame: 3, 5, and 7 minute timepoints, post-CAC on Day 1 of receiving treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 66 | 68 | 66
Units on a scale
  3 min post-CAC | 0.9 (0.8) | 2.5 (0.8) | 1.4 (0.8)
  5 min post-CAC | 1.1 (0.9) | 2.6 (0.8) | 1.5 (0.9)
  7 min post-CAC | 1.1 (0.9) | 2.5 (0.9) | 1.5 (1.0)

7. Secondary Outcome: Mean Conjunctival Redness at 24 Hours Duration of Action
Description: A treatment efficacy CAC was performed 24 hours after drop instillation. Conjunctival redness was assessed by the investigator on a 0-4 scale (0=none to 4=extremely severe). Average of conjunctival redness score over both eyes was analyzed.
Time Frame: 7, 15, and 20 minute timepoints, post-CAC on Day 1 of receiving treatment
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | AL-4943A | Vehicle | Pataday
Number analyzed (Participants) | 66 | 68 | 66
Units on a scale
  7 min post-CAC | 1.5 (0.8) | 2.1 (0.8) | 1.9 (0.8)
  15 min post-CAC | 1.8 (0.9) | 2.3 (0.7) | 2.1 (0.7)
  20 min post-CAC | 1.8 (0.9) | 2.3 (0.9) | 2.1 (0.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study. All randomized patients who received study medication were evaluable for the safety analysis.
Description: At each visit, after the patient had the opportunity to spontaneously mention any problems, the investigator inquired about adverse events by asking the standard questions: "Have you had any health problems since your last study visit?" "Have there been any changes in the medicines you take since your last study visit?"
Arm/Group | AL-4943A | Vehicle | Pataday
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/68 | 0/68
Other Adverse Events (participants affected / at risk) | 0/66 | 0/68 | 0/68

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.